CLINICAL TRIAL: NCT00493012
Title: Effects of a Vitamin D (Cholecalciferol) Supplement on Body Composition, Blood Pressure, and Lipid and Diabetes Parameters in Overweight Patients Attending a Telemedically Guided Weight Loss Program
Brief Title: Vitamin D Effects in Overweight Patients
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heart and Diabetes Center North-Rhine Westfalia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 001
Record Dates: First submitted 2007-06-26; First posted 2007-06-27 (Estimated); Results first posted 2012-03-08 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2011-05

CONDITIONS: Overweight; Obesity
Keywords: body weight; body compostion; vitamin D; blood pressure
MeSH Terms: conditions — Overweight; Obesity; Body Weight | interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- vitamin D oil (Experimental): oil containing vitamin D (Vigantol oil)
  Interventions: Dietary Supplement: vitamin D
- placebo oil (Placebo Comparator): oil not containg vitamin D (Migliol oil)
  Interventions: Dietary Supplement: vitamin D

INTERVENTIONS:
Dietary Supplement: vitamin D — 6 drops of a vitamin D containing oil

SUMMARY:
The purpose of the study is to investigate in overweight patients who are on a telemedically guided weight loss program the influence of a daily vitamin D supplement on

* weight loss and body composition,
* selected inflammation markers and biochemical parameters of lipid and glucose metabolism .
* selected clinical parameters such as blood pressure, heart rate

DETAILED DESCRIPTION:
Obese patients are known to have low levels of vitamin D metabolites. There is some evidence that vitamin D and/or dietary calcium may influence energy metabolism and body weight. We therefore perform a prospective controlled trial with 200 overweight (Body mass index 27-29.9 kg/m2) and obese subjects (Body mass index >= 30 kg/m2) who are on a telemedically guided weight loss program. Subjects randomly receive a daily vitamin D supplement or a placebo for 1 year. Participants have to send their body weight data to the study office weekly. In addition, a nutritionist at the study office has to be contacted weekly to receive further support concerning the weight loss program. Dietary records have to be completed monthly. Clinical parameters and blood samples are collected at baseline, and after 6 and 12 months. It is the aim of the study to investigate the vitamin D effects on weight loss and body composition. In addition, possible vitamin D effects on clinical and selected biochemical parameters should be assessed. These parameters include heart rate, blood pressure, inflammation markers, and parameters of lipid and glucose metablolism.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index > 27 kg/m2

Exclusion Criteria:

* pregnant and lactating women
* vegetarians
* patients with renal insufficiency (creatinine > 1.5 mg/dl)
* History of renal stones and gallstones
* patients with insulin dependent diabetes mellitus
* parallel participation in another clinical study
* missing informed consent
* subjects with pacemaker implantation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2006-01; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heinrich Koertke, MD, Principal Investigator — Institute of Applied Telemedicine, Heart and Diabetes Center North-Rhine Westfalia, 32545 Bad Oeynhausen, Germany
Locations (1):
- Heart and Diabetes Center NRW, Bad Oeynhausen, North-Rhine Westfalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zittermann A, Frisch S, Berthold HK, Gotting C, Kuhn J, Kleesiek K, Stehle P, Koertke H, Koerfer R. Vitamin D supplementation enhances the beneficial effects of weight loss on cardiovascular disease risk markers. Am J Clin Nutr. 2009 May;89(5):1321-7. doi: 10.3945/ajcn.2008.27004. Epub 2009 Mar 25. PMID 19321573
- See also: PMID: 17344484 — http://www.ncbi.nlm.nih.gov/sites/entrez
- See also: PMID: 16600341 — http://www.ncbi.nlm.nih.gov/sites/entrez
- See also: PMID: 16197570 — http://www.ncbi.nlm.nih.gov/sites/entrez

RESULTS

PARTICIPANT FLOW:
Groups:
- Experiment: A daily vitamin D supplement of 3300 IU vitamin D is given as an oily solution for 1 year.
- Placebo Comparator: A daily placebo oil is given for year
Period: Overall Study
Arm/Group | Experiment | Placebo Comparator
Started | 100 | 100
Completed | 82 | 83
Not Completed | 18 | 17
Not completed — Lost to Follow-up | 18 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Experiment | Placebo Comparator | Total
Number analyzed (Participants) | 100 | 100 | 200
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 98 | 98 | 196
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.4 (10.3) | 48.8 (10.1) | 48.1 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 72 | 134
  Male | 38 | 28 | 66
Region of Enrollment [Number; unit: participants]
  Germany | 100 | 100 | 200

OUTCOME MEASURES:

1. Primary Outcome: Change in Body Weight From Baseline to 12 Months
Time Frame: baseline, 12 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Experiment | Placebo Comparator
Number analyzed (Participants) | 82 | 83
kg | -5.7 (5.8) | -6.4 (5.6)

2. Secondary Outcome: Change in Fat Mass From Baseline to 12 Months
Time Frame: baseline, 12 months
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Experiment | Placebo Comparator
Number analyzed (Participants) | 82 | 83
kg | -4.1 (4.6) | -4.9 (4.9)

3. Secondary Outcome: Change in 25-hydroxyvitamin D From Baseline to 12 Months
Time Frame: baseline, 12 months
Measure: Mean (Standard Deviation); unit: nmol/l
Arm/Group | Experiment | Placebo Comparator
Number analyzed (Participants) | 82 | 83
nmol/l | 55.5 (55.8) | 11.8 (36.3)

4. Secondary Outcome: Change in Calcitriol From Baseline to 12 Months
Time Frame: baseline, 12 months
Measure: Mean (Standard Deviation); unit: pmol/l
Arm/Group | Experiment | Placebo Comparator
Number analyzed (Participants) | 82 | 83
pmol/l | 40.0 (95.0) | 9.3 (57.0)

5. Secondary Outcome: Change in Parathyroid Hormone From Baseline to 12 Months
Time Frame: baseline, 12 months
Measure: Mean (Standard Deviation); unit: pmol/l
Arm/Group | Experiment | Placebo Comparator
Number analyzed (Participants) | 82 | 83
pmol/l | -1.24 (2.18) | -0.91 (2.55)

6. Secondary Outcome: Change in Triglycerides From Baseline to 12 Months
Time Frame: baseline, 12 months
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Experiment | Placebo Comparator
Number analyzed (Participants) | 82 | 83
mmol/l | -0.19 (0.54) | 0.03 (0.50)

7. Secondary Outcome: Change in LDL-cholsterol From Baseline to 12 Months
Time Frame: baseline, 12 months
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Experiment | Placebo Comparator
Number analyzed (Participants) | 82 | 83
mmol/l | 0.19 (1.03) | -0.09 (0.17)

8. Secondary Outcome: Change in C-reactive Protein From Baseline to 12 Months
Time Frame: baseline, 12 months
Measure: Mean (Standard Deviation); unit: mg/l
Arm/Group | Experiment | Placebo Comparator
Number analyzed (Participants) | 82 | 83
mg/l | -0.03 (0.46) | -0.05 (0.68)

9. Secondary Outcome: Change in Tumor Necrosis Factor Alpha From Baseline to 12 Months
Time Frame: baseline, 12 months
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Experiment | Placebo Comparator
Number analyzed (Participants) | 82 | 83
pg/ml | -0.80 (2.5) | -0.26 (2.9)

10. Secondary Outcome: Change in Proinsulin From Baseline to 12 Months
Time Frame: baseline, 12 months
Measure: Mean (Standard Deviation); unit: pmol/l
Arm/Group | Experiment | Placebo Comparator
Number analyzed (Participants) | 82 | 83
pmol/l | -4.6 (14.9) | -4.1 (9.9)

11. Secondary Outcome: Change in Hb A1c From Baseline to 12 Months
Time Frame: change from baseline to 12 months
Measure: Mean (Standard Deviation); unit: % glycosylated hemoglobin
Arm/Group | Experiment | Placebo Comparator
Number analyzed (Participants) | 82 | 83
% glycosylated hemoglobin | -0.25 (0.23) | -0.25 (0.23)

ADVERSE EVENTS:
Arm/Group | Experiment | Placebo Comparator
Serious Adverse Events (participants affected / at risk) | 0/100 | 0/100
Other Adverse Events (participants affected / at risk) | 0/100 | 0/100

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes